CLINICAL TRIAL: NCT02101242
Title: Regional Cerebral Oxygen Saturation Under General Anesthesia A Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Cardiac surgery group could not be measured (technical monitoring problems)
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: ReCOSA
Record Dates: First submitted 2014-03-13; First posted 2014-04-02 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Regional Cerebral Oxygen Saturation
Keywords: Near-infrared-Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Orthopedic surgery of the shoulder: Near-infrared spectroscopy (NIRS) can detect fluctuation of regional cerebral oxygen saturation during change from supine position to beach chair position.
- Gynecological, urological or general surgery: Near-infrared spectroscopy (NIRS) can detect fluctuation of regional cerebral oxygen saturation during change from supine position to Trendelenburg position.
- Cardiac surgery: Near-infrared spectroscopy (NIRS) can detect fluctuation of regional cerebral oxygen saturation in patients undergoing cardiac surgery with cardiopulmonary bypass (heart-lung machine).

SUMMARY:
A total of 60 patients will be enrolled in the study: 20 each who receive surgery in beach chair position or Trendelenburg's position and 20 patients undergoing cardiac surgery. Regional cerebral oxygen saturation will be measured continuously during surgery. Duration and extent of deviations from individual baseline values will be recorded and detected deviations treated according to their clinically apparent cause (e.g. hypotension/hypovolaemia, anaemia, low cardiac output) in accordance with our standard operating procedures (SOPs).

Patients are then followed up until the end of hospital stay or for a maximum of 10 days after surgery. Their level of cognitive function will be tested and compared to the data acquired before surgery to detect impairment, delirium or postoperative cognitive deficit (POCD).

The purpose of this pilot study is to evaluate the design and conduct of a projected full scale observational clinical study.

DETAILED DESCRIPTION:
The primary goal of this study is the detection of perioperative fluctuations of regional cerebral oxygen saturation in patients undergoing surgery in general anaesthesia. These fluctuations will be monitored using the a non-invasive monitoring system based on the method of near-infrared spectroscopy (NIRS).

Regional cerebral hypoxia is considered one of the possible precipitating factors of postsurgical cognitive impairment (as seen in patients with postoperative cognitive deficit or postoperative delirium), but without monitoring it may easily remain undetected. A differentiated analysis of fluctuations is gained by calculation of the area under curve (AUC) of a defined deviation from individual baseline regional cerebral oxygen saturation (rSO2) over time.

When deviations are detected, they will be treated in this study according to their clinically apparent cause (e.g. hypotension/hypovolaemia, anaemia, low cardiac output) in accordance with current standard operating procedures (SOPs) to re-elevate regional cerebral oxygen saturation (rSO2) to within 20% of baseline.

Among these procedures are

1. Elevation of systemic arterial pressure by application of vasopressors
2. Consideration of systemic (pulse oxymetric) oxygen saturation
3. Adjustment of artificial ventilation subject to endexpiratory concentration of carbon dioxide (CO2)
4. Transfusion of concentrated red cells in case of Hemoglobin (Hb) <7-9 g/dl
5. Transthoracic or transesophageal echocardiogram (TTE/TEE) and assessment of centralvenous oxygen saturation in case of suspected myocardial insufficiency

which should be applied to patients of the 3 defined groups as needed.

This explorative project is a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* patients with male-to-female ratio approaching 1:1
* age ≥ 18 years
* scheduled duration of surgery longer than or equal to 60 minutes
* patients undergoing one of the following procedures:

  1. orthopedic surgery of the shoulder in beach chair position
  2. gynecological, urological or general surgery in Trendelenburg's position
  3. cardiac surgery

Exclusion Criteria:

* Moribund patients
* Persons without the capacity to consent
* Unability of German language use
* Inability of communication due to severe hearing and severe vision impairments
* Accommodation in an institution due to an official or judicial order
* Co-worker of the Charité
* Participation in another interventional study within 30 days before participation in this study
* Alcohol- use disorders according to the Alcohol Use Disorders Identification Test (AUDIT)
* Preoperative Dementia (Minimal Mental State Examination < 24)
* Stroke, traumatic brain injury within the last 12 months or patients with residual neurological deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders, over 18 years of age, undergoing elective surgery in general anesthesia.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-05-11 (Actual); Primary Completion 2014-09-14 (Actual); Study Completion 2014-09-17 (Actual)

PRIMARY OUTCOMES:
Regional cerebral oxygen saturation (rSO2) | Duration of elective surgery (an average of 2 hours)
  Regional cerebral oxygen saturation (rSO2) is measured under different body positions for elective surgery

SECONDARY OUTCOMES:
Incidence and severity of postoperative delirium | In the 10 - day postoperative sample period
  Nursing Delirium Screening Scale (Nu-DESC), Confusion Assessment Method (CAM-ICU), Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-V) (DSM-V), International Classification of Diseases (ICD)-10 (ICD-10)
Incidence and severity of postoperative cognitive dysfunction | In the 10-day postoperative sample period
  Test battery: Verbal Learning Test, Stroop Colour Word Test, Letter Digit Substitution Test, Concept Shifting Test
Rate of organ complications | In the 10-day postoperative sample period
Electrical activity of the brain | Duration of elective surgery (an average of 2 hours)
  Electrical activity of the brain is measured by electroencephalogram (EEG-derived) bispectral index (BIS) monitoring
Somatic cerebral oxygen saturation (sSO2) | Duration of elective surgery (an average of 2 hours)
  Somatic cerebral oxygen saturation (rSO2) of the lower limbs (absolutely and in side comparison) in cardiac surgery patients
Hospital length of stay | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Post-anaesthesia Discharge Scoring System (PADSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - Universitätsmedizin Berlin, Berlin, Germany